CLINICAL TRIAL: NCT03473509
Title: Impact of a Safety-Net Primary Care CKD Registry
Brief Title: Primary Care CKD Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34DK093992 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Hypertension; Chronic Kidney Diseases
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Kidney Disease (CKD) Registry (Experimental): The CKD registry provided primary care practice teams with point-of-care data about patient-specific CKD status, recent ambulatory clinic blood pressure (BP) readings, status of Angiotensin Converting Enzyme inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) prescription, and quantification of albuminuria (UACR). It also provided data about diabetes care, immunization status, and data pertinent to age appropriate cancer screening, to align with usual care. Point-of-care decision support reminded primary care providers (PCPs) about guideline concordant care for individuals with CKD. Quarterly feedback to practice teams and individual PCPs identified patients with CKD and BP >140/90 mmHg, those not prescribed an ACEi/ARB, and those with albuminuria.
  Interventions: Other: CKD Registry
- Usual Care Registry (No Intervention): Usual care consisted of an electronic registry that was in use before trial implementation. It provided practice teams with point-of-care data about diabetes care, age-appropriate cancer screening and immunizations, but no CKD-related data. Medical assistants were encouraged to use the usual care registry to identify patients who were due for cancer screening or immunizations. Quarterly feedback was not provided for practice teams randomized to receive usual care.

INTERVENTIONS:
Other: CKD Registry — Health Service intervention
  Arms: Chronic Kidney Disease (CKD) Registry

SUMMARY:
This study examines whether a safety-net primary care CKD registry directed at the entire primary care team can enhance the delivery of guideline concordant CKD care, including BP control, ACEi/ARB use and albuminuria quantification.

ELIGIBILITY:
Inclusion Criteria:

All PCPs who worked in practice teams and provided longitudinal primary care to patients were eligible to participate in this study. Practice teams that consisted of several physicians (+/- trainees), one nurse, nurse practitioners, medical assistants and behaviorists, were randomized 1:1 to one of two arms with a random number generator: access to an electronic CKD registry or a usual care registry for 12 months.

Exclusion Criteria:

PCPs who solely provided specialty care, for example HIV services or urgent care, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in clinic systolic | 12 months
  Change in ambulatory systolic BP measured at ambulatory clinic visits in the health care system.

SECONDARY OUTCOMES:
Change in proportion of patients with BP control | 12 months
  Change in the proportion of patients with BP control defined by BP <140/<90 mmHg at an ambulatory clinic visit.
Change in proportion fo patients with urine albuminuria quantification | 12 months
  Change in proportion of patients whose albuminuria was quantified by a urine test among those had not received quantification at trial initiation.
Change in albuminuria severity | 12 months
  Change in albuminuria severity (mg urine albumin/g urine creatinine) among those patients with albuminuria quantified at trial initiation
Change in proportion of patients with ACEi/ARB prescription | 12 months
  Change in proportion of patients prescribed an ACEi/ARB in the clinical record or had a documented reason for no prescription (i.e., allergy, prior development of hyperkalemia, or acute kidney injury)

IPD SHARING:
Plan to Share IPD: No
data can be shared when requested by other individual researchers